CLINICAL TRIAL: NCT06087289
Title: KANDOVA - A Two-Part Phase Ib/IIa Study to Evaluate the Safety and Tolerability of KAND567, in Combination With Carboplatin Therapy, and to Determine the Recommended Phase II Dose (RPIID) of KAND567: An Open-Label, Multicenter Dose Escalation Study With an Expansion Cohort in Women With Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: A Study to Evaluate the Safety of KAND567, in Combination With Carboplatin Therapy, in Women With Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Acronym: KANDOVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novakand Pharma AB (Industry)
Collaborators: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAN0007; 2024-515572-13-00 (EU CTIS Number); 2022-002792-11 (EudraCT Number)
Record Dates: First submitted 2023-09-27; First posted 2023-10-17 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-12

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Fractalkine; Ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Chemokine CX3CL1; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose escalation to determine Recommended Phase II Dose (RPIID) (Experimental): Part 1 of the study will include escalating doses of KAND567 administered in combination with carboplatin (according to standard of care) to approximately 10 subjects in total (may range from 6 to 24 subjects depending on DLTs). Carboplatin will be given on Day 1 of the 21-day cycle at a dose of AUC 5 according to standard of care. KAND567 will be orally administered during the first 2 weeks (Days 2 to 14) of each 21-day carboplatin cycle for up to 6 treatment cycles (or until unacceptable toxicity or disease progression).
  KAND567 dose escalation will apply for the first week (Days 2 to 7) of the treatment cycle. During the second week of the treatment cycle (Days 8 to 14), KAND567 will be administered at a fixed dose of 250 mg BID to all subjects. Doses of KAND567 will be escalated according to an adaptive, intra-individual dose escalation design.
  Interventions: Drug: KAND567; Drug: Carboplatin
- Part 2: Expansion cohort to evaluate RPIID (Experimental): An expansion cohort will be enrolled in Part 2 of the study to further evaluate the RPIID (approximately 20 subjects; may range from 6 to 24 subjects, depending on Part 1). If the number of subjects with confirmed CX3CR1 expression in tumor cells is below 50%, an additional 15 subjects may be included in Part 2 of the study.
  Carboplatin will be given on Day 1 of the 21-day cycle at a dose of AUC 5 according to standard of care. For KAND567, the RPIID will be orally administered to the cohort during the first week of each carboplatin cycle (Days 2 to 7). During the second week of the treatment cycle (Days 8 to 14), KAND567 will be administered at 250 mg BID. Up to 6 treatment cycles will be given (or until unacceptable toxicity or disease progression).
  Interventions: Drug: KAND567; Drug: Carboplatin

INTERVENTIONS:
Drug: KAND567 — KAND567 is a drug in capsule and is intended to be orally administered approximately every 12 hours (±1 hour) with an initial loading dose on Day 2 of two times the dose specified for that dose group (e.g., 2 x 250, 2 x 375, 2 x 500, or 2 x 625 mg KAND567, depending on the dose group; in Part 2, this is the RPIID), followed by a KAND567 dose (Day 2, evening dose) that corresponds to the given dose level. On Days 3 to 7, the subjects will be orally administered the specified KAND567 dose (e.g., 250, 375, 500, or 625 mg BID, depending on the dose group; in Part 2, this is the RPIID).
  During the second week of dosing (Days 8 to 14) in Part 1 and Part 2, the subjects will be orally administered KAND567 at a dose of 250 mg BID. One treatment cycle is defined as a 21-day period, and each subject will receive up to 6 treatment cycles (or until unacceptable toxicity or disease progression).
  Other Names: Fractalkine
Drug: Carboplatin — Carboplatin will be administered i.v. according to standard of care at a dose of AUC 5. One cycle is defined as a 21-day period with chemotherapy given on Day 1. Each subject will receive up to 6 treatment cycles (or until unacceptable toxicity or disease progression). The carboplatin dose should be calculated using the Calvert formula: Carboplatin dose (mg) = target AUC 5 × (GFR + 25). GFR should be calculated using the Cockcroft-Gault formula. The maximum carboplatin dose is based on a calculated GFR that is capped at 125 mL/min for subjects with normal renal function.

SUMMARY:
The study is a multicenter, Phase Ib/IIa, open-label, dose-escalation study to evaluate the safety and tolerability of orally administered KAND567 in combination with carboplatin therapy, and to determine the Recommended Phase II Dose (RPIID) of KAND567 in combination with carboplatin in subjects with recurrent platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancer.

In Part 1, dose escalation will be based on the recommendation of the Safety Review Committee (SRC) after review of the emerging safety and tolerability information. The SRC is also mandated to modify the dose levels within the dose range (125 to 625 mg BID), as well as the schedule to maintain subject safety and best serve the objectives of the study. Once the RPIID has been identified in Part 1, the SRC may recommend to the Sponsor to start Part 2.

An expansion cohort will be enrolled in Part 2 of the study to further evaluate the RPIID (approximately 20 subjects; may range from 6 to 24 subjects, depending on Part 1). If the number of subjects with confirmed CX3CR1 expression in tumor cells is below 50%, an additional 15 subjects may be included in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified high-grade serous or high-grade endometrioid epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer
* Participants* must have recurrent disease, defined as: 1st relapse 3 to 6 months after completion of the last dose of primary platinum containing treatment, or 2nd or 3rd relapse within 6 months after completion of the last dose of the latest platinum-containing regimen (platinum-free interval within 6 months)

  *Prior treatment with PARPi is allowed. In bevacizumab-naive patients, bevacizumab can be included as part of treatment after tumor progression on study drugs according to local clinical practice
* Participants must have had platinum-based chemotherapy in the first-line setting (at primary treatment or 1st relapse requiring chemotherapy)
* For BRCA status, samples must be available for analysis; for HRD status, samples should be available for analysis, if possible. If not already analyzed, the subject agrees to undergo analysis of HRD and BRCA status on primary tumor tissue and/or recurrent tumor tissue
* ECOG performance status 0-2
* Subjects must have at least 1 measurable disease according to RECIST 1.1 guidelines. Non-measurable disease must be evaluable using GCIG CA 125 criteria (CA 125 ≥ 2 x upper limit of normal [ULN]). If the subject has only 1 measurable lesion, this should not be the same lesion used for biopsy, nor should it be in a previously irradiated area.
* Able to take oral medications
* Adequate organ function: Absolute neutrophil count ≥ 1.5 x 10^9/L, Platelets > 100 x 10^9/L, Hemoglobin ≥ 80 g/dl, Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula, Total bilirubin ≤ ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ ULN
* Consent to biopsy taken prior to starting treatment and Week 8 (± 1 week) of treatment
* At least 18 years of age
* Life expectancy of at least 12 weeks
* Women of childbearing potential must use adequate birth control for the study duration and 6 months afterwards. She must use contraceptive methods with a failure rate of < 1% to prevent pregnancy* and drug exposure of a partner. Male partners must refrain from donating sperm from their partner's first IMP dose until 6 months after their partner's last IMP dose.

  * Combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD) or intrauterine hormone-releasing system (IUS); bilateral tubal occlusion, vasectomy, and sexual abstinence.
* Willingness and ability to comply with study procedures, visit schedules, study restrictions and requirements
* Able to fully understand and participate in study-related procedures, including compliance and patient reported outcome
* Written informed consent. Subjects must give informed consent prior to any study-specific procedure

Exclusion Criteria:

* Ovarian sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial cancers, and cancer types not mentioned in the inclusion criteria
* Primary platinum-refractory disease, defined as tumor progression during or within 12 weeks from end of first platinum treatment
* Concurrent cancer therapy (including anti-hormonal therapy for breast cancer unless it is omitted at the latest at study enrollment).
* Received other than platinum-containing therapy for primary disease (first-line treatment)
* Received non-platinum-containing chemotherapy line (e.g. weekly paclitaxel) in treatment of recurrent ovarian cancer. Maintenance with bevacizumab and/or PARP-inhibitor is allowed.
* Treatment with an investigational agent concurrently, or where the last dose was administered within 5 elimination half-lives or where pharmacological activity may still be present as assessed by the Investigator.
* Previous malignant disease: subjects are not eligible for the study if actively being treated for invasive cancer other than ovarian cancer. Subjects with previous malignant disease other than ovarian cancer who are relapse-free and treatment-free for more than three years may enter this study (exception: anti-hormonal therapy, which must be omitted at the latest at study enrollment). Subjects with previous history of in situ carcinoma, stage 1A cervical cancer or non-invasive basal cell and squamous cell skin carcinoma can enter this trial.
* Immunodeficiency or organ transplant. Autoimmune or inflammatory condition that requires immunosuppressive or steroid therapy during the course of the study. Subjects using immunosuppressive medications within 14 days prior to the first IMP dose, except for topical medications (intranasal, inhaled, local injection, systemic [prednisolone equivalent 10 mg/day or less]) or as needed for hypersensitivity reactions such as CT scan premedication.
* Live vaccines within 28 days prior to the first IMP dose
* Major surgery within 28 days prior to the first IMP dose, or not recovered from previous surgery to CTCAE (v5) grade 1 equivalent
* Active infection including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Transient ischemic attack (TIA) or stroke, including bleeding, within the past 6 months
* Brain metastases
* Major cardiac dysfunction defined as > NYHA II
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Serious, uncontrolled, and active infection at enrollment, as determined by the Investigator
* Pregnancy or breastfeeding
* Persistence of clinically relevant therapy-related toxicity from previous chemotherapy (≥ CTCAE grade 3, except for liver and gastrointestinal ≥ CTCAE grade 2)
* Need for concomitant use of drugs that are: moderate or strong inhibitors of CYP3A4 that may increase concentrations of KAND567; Inducers of CYP3A4 that may decrease concentrations of KAND567; highly dependent on CYP2B6, CYP2C8 or CYP3A4 for their metabolism where KAND567 may increase their concentrations. Treatment with such drugs should have been stopped at least five half-lives before initiation of KAND567 therapy. A list of drugs was provided.
* Continuous use of herbal preparations (e.g., St. John's wort) within 2 weeks prior to enrollment
* Any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (e.g., compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Known or suspected hypersensitivity to any of the IMPs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, as measured by the occurence of adverse events (AEs) | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Measured by occurence of AEs and serious adverse events (SAEs)
Evaluate the safety and tolerability of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, as measured by the occurrence of dose limiting toxicities (DLTs) | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Measured by the occurrence of DLTs
Evaluate the safety and tolerability of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, as measured by vital signs | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Measured by the occurrence of clinically abnormal vital signs
Evaluate the safety and tolerability of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, as measured by ECG | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Measured by the occurrence of clinically abnormal electrocardiography (ECG)
Evaluate the safety and tolerability of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, as measured by lab safety tests | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Measured by the occurrence of clinically abnormal lab test results (routine clinical chemistry, haematology, and urinalysis)
Determine the Recommended Phase II Dose (RPIID) of KAND567 in combination with carboplatin therapy in recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer | From the first KAND567 IMP administration to the subject (Day 2) until the end of study visit (Week 20).
  In Part 1/Phase Ib, RPIID of KAND567 in combination with carboplatin therapy will be determined based on safety and tolerability (DLTs).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Week 12 and 18
  Evaluate ORR according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Gynecologic Cancer Intergroup (GCIG) definitions, i.e., best overall response in subjects with measurable disease, or without measurable disease who are evaluable by CA 125.
Progression-Free Survival (PFS) | From the first IMP administration to the subject (Day 1) to Week 12 and 18
  Evaluate PFS according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Gynecologic Cancer Intergroup (GCIG) definitions, i.e., the time from start of treatment to disease progression or death.
Overall survival (OS) | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Evaluate OS according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Gynecologic Cancer Intergroup (GCIG) definitions, i.e., the time from the start of treatment to death due to any cause.
Disease control rate (DCR) | Week 12 and 18
  Evaluate DCR, i.e., Complete response (CR) + Partial response (PR) + Stable disease (SD), according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Gynecologic Cancer Intergroup (GCIG) definitions, where: CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameter; and SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Duration of response | From the first IMP administration to the subject (Day 1) until the end of study visit (Week 20)
  Evaluate duration of response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Gynecologic Cancer Intergroup (GCIG) definitions, i.e., time from documentation of tumor response to disease progression.
Change in pain score | From baseline (Week 1) to Weeks 4, 7, 10, 13, 16 and 20.
  Change in pain score (patient reported outcome), as measured by the Numeric Rating Scale (NRS). The NRS is a scale rating pain from "no pain" to "worst pain possible" from 0 to 10, where a higher value indicates greater pain intensity.
Determine the plasma exposure of KAND567 | For each 21-day treatment cycle, on Day 7 (0, 1, 2, and 4 hours after KAND567 morning dose) and Day 14 (0, 2 and 4 hours after KAND567 morning dose). Each subject receives up to 6 treatment cycles (or until unacceptable toxicity or disease progression)
  Blood samples will be collected for the determination of concentrations of KAND567 in plasma. The determination of the total concentration of KAND567 in plasma will be carried out using Liquid Chromatography - Tandem Mass Spectrometry (LC-MS/MS). KAND567 PK drug concentration data will be graphically visualized together with normalized PK drug concentration data from the previous KAN0001 study (i.e., no formal PK analysis will be performed).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Dahlstrand, MD/PhD, Principal Investigator — Karolinska University Hospital
Locations (4):
- Odense University Hospital, Odense, Denmark
- Oslo University Hospital, Oslo, Norway
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Solna

IPD SHARING:
Plan to Share IPD: No